CLINICAL TRIAL: NCT00043082
Title: A Phase III Study of Liposomal Doxorubicin Plus Carboplatin Versus Carboplatin in Platinum-Sensitive Patients With Recurrent Epithelial Ovarian and Peritoneal Carcinoma After Failure of Initial Platinum-Based Chemotherapy
Brief Title: S0200 Carboplatin With or Without Doxil in Patients With Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000256331; S0200 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2002-08-05; First posted 2003-01-27 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: peritoneal cavity cancer; recurrent ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- carboplatin and doxorubicin (Experimental): carboplatin and liposomal doxorubicin given q 4 weeks
  Interventions: Drug: carboplatin; Drug: pegylated liposomal doxorubicin hydrochloride
- carboplatin (Active Comparator): carboplatin alone
  Interventions: Drug: carboplatin

INTERVENTIONS:
Drug: carboplatin — intravenous q 4 weeks
Drug: pegylated liposomal doxorubicin hydrochloride — intravenous q 4 weeks
  Arms: carboplatin and doxorubicin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known if carboplatin is more effective with or without liposomal doxorubicin in treating recurrent ovarian epithelial or primary peritoneal cancer.

PURPOSE: Randomized phase III trial to determine the effectiveness of carboplatin with or without liposomal doxorubicin in treating patients who have recurrent ovarian epithelial or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare overall survival of patients with platinum-sensitive recurrent ovarian epithelial or primary peritoneal cancer treated with carboplatin with or without pegylated doxorubicin HCl liposome.
* Compare progression-free survival, confirmed complete response rates, and time to treatment failure in patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to disease measurability (elevated CA 125 only vs nonmeasurable disease only with or without elevated CA 125 vs measurable disease), number of disease sites (2 or fewer vs 3 or more), and serous tumor histology (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive carboplatin IV over 15 minutes and pegylated doxorubicin HCl liposome IV over 1 hour on day 1.
* Arm II: Patients receive carboplatin IV as in arm I. Treatment in both arms repeats every 4 weeks for a total of 15 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed at 4 weeks, every 6 months for 3 years, and then annually for 7 years.

PROJECTED ACCRUAL: A total of 900 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial carcinoma

  * Stage III or IV disease at time of initial staging laparotomy
* Primary peritoneal and mixed Mullerian tumors allowed
* No borderline ovarian tumors
* Disease progression or recurrence after a progression-free and platinum-free interval of 6-24 months after completion of first-line platinum-based chemotherapy (either single agent or combination therapy)
* Disease progression or recurrence based solely on CA 125 elevation allowed, provided that one of the following is true:

  * Prior baseline CA 125 greater than 35 U/mL and subsequent normalization of no greater than 35 U/mL must have CA 125 greater than 2 times upper limit of normal (ULN) on 2 occasions at least 1 week apart
  * Prior baseline CA 125 greater than 35 U/mL that never normalized must have CA 125 greater than 2 times the nadir value on 2 occasions at least 1 week apart
  * Prior normal baseline CA 125 (no greater than 35 U/mL) must show CA 125 greater than 2 times ULN on 2 occasions at least 1 week apart
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic

* SGOT and/or SGPT no greater than 2 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2 times ULN
* Bilirubin no greater than ULN

Renal

* Creatinine no greater than 1.9 mg/dL

Cardiovascular

* No New York Heart Association class II-IV cardiac disease
* No clinical evidence of congestive heart failure
* Ejection fraction greater than 50% by MUGA or 2-dimensional echocardiogram

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or incidental carcinoid cancer
* No evidence of active or uncontrolled infection
* No severe gastrointestinal symptoms (i.e., partial obstruction) and/or gastrointestinal bleeding or diarrhea
* No greater than grade 1 preexisting sensory neuropathy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 28 days since prior biologic consolidation therapy
* No concurrent immunotherapy

Chemotherapy

* See Disease Characteristics
* At least 28 days since prior non-platinum-containing consolidation chemotherapy
* No prior pegylated doxorubicin HCl liposome
* No prior cumulative anthracycline (e.g., doxorubicin, daunorubicin, epirubicin) dose in excess of 240 mg/m^2
* No other concurrent chemotherapy

Endocrine therapy

* No concurrent hormonal therapy

Radiotherapy

* No prior abdominopelvic irradiation
* No concurrent radiotherapy

Surgery

* See Disease Characteristics
* At least 28 days since prior surgical debulking for disease progression or recurrence and recovered
* No concurrent surgery

Other

* No other prior treatment during the 6-24 month progression-free and platinum-free interval except up to 12 courses of consolidation therapy
* No other concurrent anticancer therapy

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2002-08; Primary Completion 2007-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
overall survival | ten years
  From date of registration to date of death

SECONDARY OUTCOMES:
progression free survival and response | 10 years
  response by RECIST criteria
side effects | 15 months
  side effects described per NCI CTC version 2.0

CONTACTS AND LOCATIONS:
Overall Officials: David S. Alberts, MD, Study Chair — University of Arizona
Locations (91):
- United States (91):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Carl T. Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - California Cancer Center at Woodward Park Office, Fresno, California
  - Veterans Affairs Medical Center - Loma Linda (Pettis), Loma Linda, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Cancer Center, Orange, California
  - University of California Davis Cancer Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - MBCCOP - Howard University Cancer Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Health System, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield, Southfield, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Hospital Cancer Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - University of Tennessee Cancer Institute at Methodist Central Hospital, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Veterans Affairs Medical Center - Amarillo, Amarillo, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - Puget Sound Oncology Consortium, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington

REFERENCES:
- [Result] Alberts DS, Liu PY, Wilczynski SP, Clouser MC, Lopez AM, Michelin DP, Lanzotti VJ, Markman M; Southwest Oncology Group. Randomized trial of pegylated liposomal doxorubicin (PLD) plus carboplatin versus carboplatin in platinum-sensitive (PS) patients with recurrent epithelial ovarian or peritoneal carcinoma after failure of initial platinum-based chemotherapy (Southwest Oncology Group Protocol S0200). Gynecol Oncol. 2008 Jan;108(1):90-4. doi: 10.1016/j.ygyno.2007.08.075. Epub 2007 Oct 18. PMID 17949799
- [Derived] Newhouse R, Nelissen E, El-Shakankery KH, Rogozinska E, Bain E, Veiga S, Morrison J. Pegylated liposomal doxorubicin for relapsed epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Jul 5;7(7):CD006910. doi: 10.1002/14651858.CD006910.pub3. PMID 37407274